CLINICAL TRIAL: NCT06885034
Title: A Phase 1b/2, Multicenter, Open-label Study to Evaluate the Efficacy and Safety of GSK5764227 Alone and in Combination in Participants With Previously Treated Advanced Unresectable or Metastatic Gastrointestinal Solid Tumors
Brief Title: A Study to Test the Safety and Effectiveness of GSK5764227, Alone or With Other Treatments, in Participants With Advanced Gastrointestinal Cancers That Cannot be Surgically Removed
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 223675; 2025-520672-26 (Other: EU CTR)
Record Dates: First submitted 2025-03-13; First posted 2025-03-19 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Gastrointestinal Neoplasms
Keywords: GSK5764227; Solid Tumors; Colorectal Cancer; Pancreatic ductal adenocarcinoma
MeSH Terms: conditions — Gastrointestinal Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- CRC-A: GSK5764227 (Dose 1) (Experimental)
  Interventions: Biological: GSK5764227
- CRC-A: GSK5764227 (Dose 2) (Experimental)
  Interventions: Biological: GSK5764227
- CRC-B: GSK5764227 (Dose 3) (Experimental)
  Interventions: Biological: GSK5764227
- CRC-B: GSK5764227 (Dose 4) (Experimental)
  Interventions: Biological: GSK5764227
- PDAC: GSK5764227 (Dose 5) (Experimental)
  Interventions: Biological: GSK5764227

INTERVENTIONS:
Biological: GSK5764227 — GSK5764227 will be administered

SUMMARY:
This study will check how well a new medicine, GSK5764227, works, how safe it is and how the body handles it in participants all around the world with advanced inoperable or metastatic gastrointestinal cancer who have previously received treatment.

ELIGIBILITY:
Inclusion criteria:

Participants are eligible to be included in the study only if all of the following criteria apply:

• Is at least 18 or the legal age of consent in the jurisdiction in which the study is taking place years of age at the time of signing the informed consent form (ICF).

CRC Cohort

* Has histologically confirmed unresectable/, locally advanced or unresectable metastatic adenocarcinoma of the colon or rectum (histology defined by World Health Organization (WHO) classification).
* Must have received at least 1 and no more than 2 lines of systemic treatment for advanced colorectal cancer (CRC), with documented progression on most recent prior line of therapy.
* Must provide tumor tissue from a newly obtained fresh biopsy or an archival tumor tissue.

PDAC Cohort

* Has histologically or cytologically confirmed unresectable, locally advanced or metastatic adenocarcinoma of the pancreas (histology defined by WHO classification).
* Must have received 1 and no more than 1 line of therapy for advanced PDAC, with documented progression.
* Should provide tumor tissue at screening, where available or medically feasible.

All Cohorts

* Has at least 1 target lesion per RECIST 1.1, as determined by the investigator.
* Is willing to use adequate contraception.
* Is capable of giving signed informed consent, including compliance with the requirements and restrictions listed in the ICF and in the protocol.
* Has an ECOG performance status of 0 or 1.
* Has adequate organ function.

Exclusion criteria:

Participants are excluded from the study if any of the following criteria apply:

* Has a malignancy (except disease under study) that has progressed or required active treatment within the past 24 months except for basal cell or squamous cell carcinomas of the skin or in-situ carcinomas [e.g., breast, cervix, bladder] that have been resected with no evidence of disease.
* Has had any major surgery within 28 days prior to randomization (CRC Cohort) or first dose of study intervention (PDAC Cohort).
* Has any history of prior allogenic or autologous bone marrow transplant or other solid organ transplant.
* Has known sensitivity to study intervention components or excipients or other allergy that, in the opinion of the investigator or medical monitor, contraindicates participation in the study.
* Has severe, uncontrolled or active cardiovascular disorders.
* Has serious or poorly controlled hypertension.
* Has clinically significant bleeding symptoms or significant bleeding tendency within 1 month prior to the first dose.
* Has serious infection within 4 weeks prior to the first dose.
* Known active infectious diseases requiring systemic treatment or known Human immunodeficiency virus (HIV).
* Has serious arteriovenous thromboembolic events (such as deep vein thrombosis, pulmonary embolism, etc.) within 3 months prior to the first dose.
* Has untreated brain or Central nervous system (CNS) metastases or brain/CNS metastases that have progressed.
* Has current active pneumonitis or any history of pneumonitis requiring steroids or immunomodulatory treatment within 90 days of planned [randomization] or any history of drug-induced pneumonitis.
* Has a history of autoimmune disease that has required systemic treatments in the 2 years prior to screening.
* Has any active renal condition (e.g., infection, requirement for dialysis, or any other significant renal condition that could affect the participant's safety).
* Has ongoing adverse reaction(s) from prior therapy that has(have) not recovered to Grade 1 or to the baseline status preceding prior therapy.
* Has any serious and/or unstable medical or psychiatric disorder or other condition(s) (including laboratory assessment abnormalities) that could interfere with the participant's safety, obtainment of informed consent, or compliance to the study procedures.
* Has cirrhosis or current unstable liver or biliary disease per investigator assessment defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal/gastric varices, or persistent jaundice.
* Has documented presence of Hepatitis B surface antigen (HBsAg) or HBcAb at screening or within 3 months prior to the first dose of study intervention.
* Has a positive Hepatitis C virus (HCV) antibody test result at screening or within 3 months prior to the first dose of study intervention.
* Has a positive HCV RNA test result at screening or within 3 months prior to the first dose of study intervention.
* Has received immunosuppressive agents within 30 days prior to first dose of study intervention (or requires long-term [30 days or longer]).
* Has received any prior therapy with an Antibody-drug conjugate (ADC) with a Topoisomerase-1 (TOPO1)-inhibitor payload.
* Has received any live vaccine within 30 days of randomization (CRC Cohort) or before first dose of study intervention (PDAC Cohort).
* Is currently enrolled or has participated in any other clinical study involving an investigational study intervention or any other type of interventional medical research and/or has received treatment with any anticancer or investigational agent within 4 weeks prior to randomization.
* Is pregnant or breastfeeding.
* Is unable to adhere to the protocol defined SoA, including requirements for the Follow-up Period of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2025-06-11 (Actual); Primary Completion 2027-11-11 (Estimated); Study Completion 2028-06-23 (Estimated)

PRIMARY OUTCOMES:
Confirmed Objective Response Rate (ORR) | Up to approximately 22 months
  Confirmed ORR is defined as the proportion of participants who have achieved best overall response (BOR) of confirmed complete response (CR) or partial response (PR) as assessed by investigator, according to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1)

SECONDARY OUTCOMES:
Unconfirmed ORR | Up to approximately 37 months
  Unconfirmed ORR is defined as the proportion of participants who have achieved a BOR of CR or PR as assessed by investigator, according to RECIST 1.1.
Duration of Response (DoR) | Up to approximately 37 months
  DoR is defined as the time from the date of the first documented objective response (CR/PR as assessed by investigator according to RECIST 1.1) until the date of the first documented progressive disease (PD) or death, whichever is earlier.
Progression Free Survival (PFS) | Up to approximately 37 months
  PFS (assessed by investigator), defined as the time from date of randomization (for participants in CRC-A and CRC-B) or the date of first dose study intervention for participants in PDAC until the earliest date of documented disease progression per RECIST 1.1 or death due to any cause.
Number of participants with AEs, serious adverse events (SAEs) and adverse events of special interest (AESIs) by severity | Up to approximately 37 months
Number of participants with AEs leading to dose modifications, discontinuation of study interventions or death | Up to approximately 37 months
Changes from baseline in vital signs: Temperature (degree Celsius) | Baseline (Day 1) and up to approximately 37 months
Changes from baseline vital signs: Respiratory rate (breaths per minute) | Baseline (Day 1) and up to approximately 37 months
Changes from baseline vital signs: Pulse rate (beats per minute) | Baseline (Day 1) and up to approximately 37 months
Changes from baseline vital signs: Blood pressure [millimetres of mercury (mmHg) | Baseline (Day 1) and up to approximately 37 months
Changes from baseline in hematology parameters: [White blood cell count (WBCs per microliter) | Baseline (Day 1) and up to approximately 37 months
Changes from baseline in hematology parameters: [Haemoglobin (Hgb) (grams per deciliter) | Baseline (Day 1) and up to approximately 37 months
Changes from baseline in hematology parameters:[Haematocrit (Proportion of red blood cells in blood) | Baseline (Day 1) and up to approximately 37 months
Changes from Baseline haematology parameter: [Red Blood Cell Count (RBC) (million cells per microliter) | Baseline (Day 1) and up to approximately 37 months
Changes from baseline haematology parameters: Neutrophils, Lymphocytes, Monocytes, Eosinophils, Basophils (giga cells per liter) | Baseline (Day 1) and up to approximately 37 months
Changes from Baseline haematology parameter: Platelet count (cells per microliter) | Baseline (Day 1) and up to approximately 37 months
Changes from baseline Clinical chemistry parameters: Total Protein, Albumin (Grams per deciliter) | Baseline (Day 1) and up to approximately 37 months
Changes from baseline Clinical Chemistry parameters: AST/SGOT, ALT/ SGPT, ALP and CPK (International Units per liter) | Baseline (Day 1) and up to approximately 37 months
  Clinical chemistry parameters such as Aspartate Aminotransferase (AST) / Serum Glutamic-Oxaloacetic Transaminase (SGOT), Alanine Aminotransferase (ALT)/ Serum Glutamic-Pyruvic Transaminase and (SGPT), Alkaline phosphatase (ALP) and Creatinine Phosphokinase (CPK) will be analysed
Changes from baseline Clinical Chemistry parameters: Total Bilirubin and Direct Bilirubin, Glucose, Calcium, Potassium, Sodium, Magnesium, Urea Nitrogen or urea, and Creatinine (milligrams per deciliter) | Baseline (Day 1) and up to approximately 37 months
Changes from baseline Clinical Chemistry parameters: Lactate dehydrogenase, Amylase and Lipase (units per liter) | Baseline (Day 1) and up to approximately 37 months
Changes from baseline Clinical Chemistry parameters: Chloride (millimoles per liter) | Baseline (Day 1) and up to approximately 37 months
Changes from baseline Clinical Chemistry parameters: Creatinine clearance (milliliters per minute) | Baseline (Day 1) and up to approximately 37 months
Changes from baseline cardiac function: Electrocardiogram (ECG) (milliseconds) | Baseline (Day 1) and up to approximately 37 months
Changes from baseline Eastern Cooperative Oncology Group performance status (ECOG-PS) | Baseline (Day 1) and up to approximately 37 months
Maximum observed concentration (Cmax) of GSK5764227 (conjugated antibody) and GSK5757810 (small molecule toxin) | Up to approximately 37 months
Time to reach Cmax (Tmax) of GSK5764227 (conjugated antibody) and GSK5757810 (small molecule toxin) | Up to approximately 37 months
Area under the concentration-time curve (AUC) of GSK5764227 (conjugated antibody) and GSK5757810 (small molecule toxin) | Up to approximately 37 months
Number of participants with Antidrug antibody (ADA) or Neutralizing Antibody (NAb) | Up to approximately 37 months
Titers of ADA against GSK5764227 | Up to approximately 37 months
Number of participants with symptomatic AEs, by severity, as measured by Patient Reported Outcomes Version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE) | Up to approximately 37 months
  The PRO-CTCAE is a patient-reported outcome measure developed to evaluate symptomatic toxicity in participants on cancer clinical trials. The PRO-CTCAE includes a library of 124 items representing 78 symptomatic toxicities drawn from the CTCAE
Level of bother of AEs as measured by Functional Assessment of Cancer Therapy - Item GP5 (FACT-GP5) | Up to approximately 37 months
  The FACT-GP5 item is a single item from the FACT-G that assesses how bothersome the side effects of treatment are for cancer patients. The item has a 5-category response scale ranging from 0 to 4. Higher scores indicate a higher degree of AE bother.

CONTACTS AND LOCATIONS:
Locations (41):
- United States (7):
  - GSK Investigational Site, Los Alamitos, California
  - GSK Investigational Site, Whittier, California
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Durham, North Carolina
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Wenatchee, Washington
- Australia (2):
  - GSK Investigational Site, Heidelberg, Victoria
  - GSK Investigational Site, Melbourne, Victoria
- Belgium (4):
  - GSK Investigational Site, Bonheiden
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Leuven
  - GSK Investigational Site, Roeselare
- Brazil (3):
  - GSK Investigational Site, Porto Alegre
  - GSK Investigational Site, São Paulo
  - GSK Investigational Site, Teresina
- Canada (2):
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Sherbrooke, Quebec
- France (2):
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Villejuif
- GSK Investigational Site, Pisa, Italy
- Japan (5):
  - GSK Investigational Site, Aichi
  - GSK Investigational Site, Chiba
  - GSK Investigational Site, Hokkaido
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Tokyo
- Netherlands (2):
  - GSK Investigational Site, Amsterdam
  - GSK Investigational Site, Utrecht
- Norway (3):
  - GSK Investigational Site, Lrenskog
  - GSK Investigational Site, Oslo
  - GSK Investigational Site, Stavanger
- Poland (2):
  - GSK Investigational Site, Brzozów
  - GSK Investigational Site, Warsaw
- GSK Investigational Site, Seoul, South Korea
- Spain (5):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Pamplona
  - GSK Investigational Site, Santander
  - GSK Investigational Site, Zaragoza
- Sweden (2):
  - GSK Investigational Site, Lund
  - GSK Investigational Site, Stockholm

IPD SHARING:
Plan to Share IPD: Yes
Study Sponsor will assess requests from qualified researchers for anonymized individual patient-level data and related study documents. Data sharing is subject to certain criteria, conditions, and exceptions. For further information, refer to https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or asset(s) with development terminated across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months, but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf